CLINICAL TRIAL: NCT06043609
Title: Outcome Evaluation After Fertility Preservation
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2023.346
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Fertility Issues
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When patients come back after the use of frozen gametes, embryos or tissue, discarded or residual cryopreserved gamete, embryos or tissue will be used for histological and pathological assessment to determine its quality. Donated samples cannot be retrieved/ used for future fertility treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational cohort study — This is an observational cohort study

SUMMARY:
It is important to evaluate outcomes after different fertility preservation strategies. Therefore, this study aims to assess the outcomes after different fertility preservation strategies and identify any factors that may affect their reproductive outcome.

DETAILED DESCRIPTION:
All patients who have undergone or will seek fertility preservation services in PWH will be invited to participate. For those patients who have undergone fertility preservation services in PWH, when they come back to use their frozen gametes or embryos, they will also be invited to participate.

Medical record assessment When patients come for fertility preservation consultation in PWH, they will be invited to participate. The medical notes of these patients undergoing fertility preservation services will be reviewed. The baseline characteristics including the socio-demographic background, past medical history, details of the surgical procedures, and the subsequent reproductive outcome, will be obtained by reviewing their hospital record. The participants will not be required to take any extra procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 0-50 years old
* Patients with any illness or who will undergo any type of treatment that may cause irreversible damage to their fertility, such as extensive abdominal surgery, high toxicity medication and treatments;
* Patients seek for fertility preservation services

Exclusion Criteria:

-Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who have undergone or will seek for fertility preservation services in PWH will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2033-10-01 (Estimated); Study Completion 2035-10-01 (Estimated)

PRIMARY OUTCOMES:
To determine any factors that may affect the success rate of different fertility preservation methods. | 10 years
  The medical notes of these patients undergoing fertility preservation services will be reviewed. The baseline characteristics including the socio-demographic background will be obtained by reviewing their hospital record.

SECONDARY OUTCOMES:
To assess the pregnancy rate after different fertility preservation methods. | 10 years
  The medical notes of these patients undergoing fertility preservation services will be reviewed. The subsequent reproductive outcome will be obtained by reviewing their hospital record.
To report on the frequency of surgical complications | 10 years
  The medical notes of these patients undergoing fertility preservation services will be reviewed. The details of the surgical procedures will be obtained by reviewing their hospital record.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline CHUNG, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No